CLINICAL TRIAL: NCT05243485
Title: Prehospital Triage of Patients With Suspected Non-ST-segment Elevation Acute Coronary Syndrome: the TRIAGE-ACS Study
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Pieter-Jan Vlaar, Principal investigator, Catharina Ziekenhuis Eindhoven
Other Study IDs: TRIAGE ACS
Record Dates: First submitted 2022-01-26; First posted 2022-02-17 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: ACS; NSTEMI - Non-ST Segment Elevation MI; Unstable Angina
Keywords: Prehospital; Risk stratification; Triage; Emergency Medical Services
MeSH Terms: conditions — Non-ST Elevated Myocardial Infarction; Angina, Unstable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1 (reference group): 500 patients will be included as an observatory control group and as a reference group to the second cohort. The PreHEART score is calculated without further consequences for triage in the ambulance and are transferred to the ED of the nearest hospital for standard care.
- Cohort 2 (intervention group): 500 patients will be included in the interventional cohort. The calculated PreHEART score has consequences for triage in the ambulance. If the PreHEART score is ≥ 5, the patient is classified as a high-risk patient for having NSTE-ACS. These patients are immediately transferred to the ED of the nearest PCI center for further diagnostic examination and to rule out other life-threatening pathologies. When the PreHEART score is ≤ 4, the patient is classified as a low-risk patient for having NSTE-ACS and is transferred to the ED of the nearest hospital without PCI facilities (non-PCI center) for further diagnostic work-up
  Interventions: Diagnostic Test: PreHEART

INTERVENTIONS:
Diagnostic Test: PreHEART — The PreHEART score is validated for use in the pre-hospital setting.The score can be calculated based on five different elements: history, ECG, age, gender, and a Point-of-Care (POC)-Troponin. A minimum of 0 points and a maximum of 2 points can be scored in each element, the total PreHEART can contain a maximum of 10 points. The score of the history is based on the symptoms of the patient in accordance with the symptoms of a myocardial infarction. Based on the suspicion of ischemia on the ECG. Age will be based on the date of birth. Compared to the female gender, the male gender has higher risk of developing myocardial infarction and will be scored higher. The biomarker Troponin will be collected via intravenous access and measured using a POC-analyzer "I-Stat" from Abbott industries. In total 17 µl of blood is required to fill a cardiac Troponin I (cTnI) cartridge. Analyzing the blood will take approximately 10 minutes.
  Groups: Cohort 2 (intervention group)

SUMMARY:
With the Emergency Medical Services (EMS), no prehospital risk stratification and triage is performed for patients suspected of having an Non-ST-segment elevation Acute Coronary Syndrome (NSTE-ACS). While the latest ESC Guidelines recommend an early invasive strategy within 24 hours for all high risk NSTE-ACS patients and same-day transfer to a PCI (Percutaneous Coronary Intervention) center. With the potential emerging logistical problem surrounding this, prehospital risk stratification and triage can have great benefits in this population as well, especially in patients with a high risk of having an NSTE-ACS. The recently validated PreHEART score makes it possible to stratify patients in a low-risk and high-risk group for having a NSTE-ACS and gives the EMS the opportunity to make triage decisions in the prehospital setting. Patients with a high risk for having an NSTE-ACS are transferred directly to an PCI-center for further diagnostic work-up. Patients with a low risk for having NSTE-ACS and transferred to the ED of the nearest hospital without PCI facilities (non-PCI center) for further diagnostic work-up, resulting in an optimization of the regional care utilization.

This is the first study to focus on patients who are at a high risk of having an NSTE-ACS and to assess if whether prehospital triage using the PreHEART score is able to significantly reduce time to final invasive diagnostics and revascularization in patients in need of coronary revascularization.

ELIGIBILITY:
Inclusion Criteria:

* Chest pain suspected for NSTE-ACS
* Age ≥ 18 years
* Intention to transfer patient to Emergency Department

Exclusion Criteria:

* ST-segment elevation Acute Coronary Syndrome
* Post resuscitation patients
* Hemodynamic instability defined as Killip Class IV
* Suspected other life treating pathology
* Pregnancy
* No informed consent for data usage

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suspected for NSTE-ACS presenting in the prehospital setting with the EMS
Sampling Method: Probability Sample
Enrollment: 1071 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-12-19 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Time from first medical contact to final invasive diagnostics and revascularization | Time from first medical contact by EMS to final invasive diagnostics and revascularization, up to 60 days
  Duration of time from first medical contact (in the EMS) to final invasive diagnostics and revascularization

SECONDARY OUTCOMES:
Number of participants with ischemic complications | 2 years
  Refractory ischemia, new myocardial infarction
Logistics during hospitalization | 30 days
  Time from first medical contact to invasive diagnostics Time from invasive diagnostics to revascularization Time from first medical contact to revascularization Duration of hospital admission Number of invasive procedures Numbers of transfers between hospitals by EMS services
Number of participants with Major Adverse Cardiac Events | 7 and 30 days
  All cause death Myocardial infarction Revascularization Stroke
Number of participants who suffer all cause death | 1 and 2 years
  Death from any cause
Number of participants with safety endpoints during invasive diagnostics and/or revascularization | During hospitalization, up to 60 days
  Bleeding complications Contrast-induced nefropathy Possible or definite stent thrombosis Ischemic stroke Death
Economic endpoints | During hospitalization, up to 60 days
  Total costs per patient stratified to low- and high-risk groups

CONTACTS AND LOCATIONS:
Locations (1):
- Catharina Hospital, Eindhoven, North Brabant, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Sagel D, Vlaar PJ, van Roosmalen R, Waardenburg I, Nieuwland W, Lettinga R, van Barneveld R, Jorna E, Kijlstra R, van Well C, Oomen A, Bartels L, Anthonio R, Hagens V, Hofma S, Gu Y, Drenth D, Addink R, van Asselt T, van der Meer P, Lipsic E, Juarez Orozco L, van der Harst P. Prehospital risk stratification in patients with chest pain. Emerg Med J. 2021 Nov;38(11):814-819. doi: 10.1136/emermed-2020-210212. Epub 2021 Aug 9. PMID 34373266
- [Derived] Demandt JPA, Koks A, Sagel D, Haest R, Heijmen E, Thijssen E, El Farissi M, Eerdekens R, van der Harst P, van 't Veer M, Dekker L, Tonino P, Vlaar PJ. External validation of the preHEART score and comparison with current clinical risk scores for prehospital risk assessment in patients with suspected NSTE-ACS. Emerg Med J. 2024 Sep 25;41(10):610-616. doi: 10.1136/emermed-2023-213866. PMID 39074964
- [Derived] Demandt J, Koks A, Sagel D, van Hattem VAE, Haest RJ, Heijmen E, Thijssen H, Otterspoor LC, van Veghel D, Eerdekens R, El Farissi M, Teeuwen K, Wijnbergen I, van der Harst P, Pijls NHJ, van 't Veer M, Tonino PAL, Dekker LRC, Vlaar PJ. Prehospital risk assessment and direct transfer to a percutaneous coronary intervention centre in suspected acute coronary syndrome. Heart. 2024 Feb 23;110(6):408-415. doi: 10.1136/heartjnl-2023-323346. PMID 38040452